CLINICAL TRIAL: NCT01836497
Title: SD01 Master Study (Safety and Efficacy Study)
Status: Completed | Type: Observational
Sponsor: Biotronik SE & Co. KG (Industry)
Responsible Party: Sponsor
Other Study IDs: TA103
Record Dates: First submitted 2013-04-12; First posted 2013-04-22 (Estimated); Last update posted 2025-01-22 (Actual); Status verified 2024-07

CONDITIONS: Ventricular Tachycardia; Ventricular Fibrillation; Heart Failure
MeSH Terms: conditions — Tachycardia, Ventricular; Ventricular Fibrillation; Heart Failure

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: SD01 ICD lead

SUMMARY:
The study is designed to confirm safety and efficacy of the SD01 ICD (implantable cardioverter-defibrillator) lead.

ELIGIBILITY:
Inclusion Criteria:

* Standard indication for an ICD/CRT-D therapy
* Signed informed consent form
* Patient is willing and able to participate for the whole study duration
* Patient is willing and able to activate and use the CardioMessenger
* Legal capacity and ability to consent.

Exclusion Criteria:

* Standard contraindication for an ICD/CRT-D therapy
* Age <18 years.
* Pregnant or breastfeeding
* Cardiac surgery is planned within the next six months
* Any condition that in the opinion of the investigator would preclude compliance with the study protocol during the whole follow-up period
* Enrollment in another cardiac clinical investigation with active treatment arm
* Mechanical tricuspid valve prosthesis or severe tricuspid valve disease
* Dexamethasone acetate intolerance

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with standard ICD/CRT-D (cardiac resynchronization therapy plus defibrillator) indication
Sampling Method: Non-Probability Sample
Enrollment: 163 (Actual)
Dates: Start 2013-05; Primary Completion 2014-12-22 (Actual); Study Completion 2024-09-25 (Actual)

PRIMARY OUTCOMES:
Rate of appropriate sensing and pacing | at the 3-month follow-up
  The evaluation of right ventricular sensing performance is based on the assessment of consecutive intrinsic beats documented with markers on an IEGM (intra-cardiac electrogram). The evaluation of ventricular sensing performance is based on the data to be collected during the 3-month follow-up. The appropriate pacing performance in the right ventricle results from the evaluation of "capture" at the end of the 3-month follow-up.
Serious adverse device effects (SADEs) related to the SD01 lead | until the 3-month follow-up

SECONDARY OUTCOMES:
Comparison of pacing threshold between Linoxsmart and SD01 | at the 3-month follow-up
  Comparison of the manually measured pacing threshold of the SD01 lead system to the Linox SD lead at 3-month follow-up. The idea is that the pacing threshold will be similar within a suitable range.
Shift rate of the painless shock impedance measurement | between 3- and 6-month follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Roland Richard Tilz, Prof. Dr. med., Principal Investigator — University Clinic of Schleswig-Holstein, Lübeck, Germany
Locations (14):
- St. Ann University Hospital, Brno, Czechia
- France (2):
  - CHU de Saint-Etienne, Saint-Etienne
  - Hopital Civil Strasbourg, Strasbourg
- Germany (8):
  - Helios Klinik Aue, Aue
  - Universitätsklinikum Düsseldorf, Düsseldorf
  - Universitätsklinik Jena, Jena
  - University Clinic of Schleswig-Holstein, Lübeck
  - Carl-von-Basedow Clinic, Merseburg
  - Städtisches Klinikum München Bogenhausen, München
  - Klinik Rothenburg, Rothenburg upon Tauber
  - Universitätsklinik Würzburg, Würzburg
- Hungary (2):
  - Semmelweiss University Hospital, Budapest
  - University of Debrecen, Debrecen
- Bovas P. Stradina KUS Latvian Center of Cardiology, Riga, Latvia